CLINICAL TRIAL: NCT03020030
Title: Treatment of Newly Diagnosed Acute Lymphoblastic Leukemia in Children and Adolescents
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Servier (Industry)
Responsible Party: Principal Investigator, Melissa Burns, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-001
Record Dates: First submitted 2017-01-06; First posted 2017-01-13 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Acute Lymphoblastic Leukemia, Pediatric
Keywords: acute lymphoblastic leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — pegaspargase; asparaginase erwinia chrysanthemi recombinant; Asparaginase; Cyclophosphamide; Cytarabine; Dasatinib; Dexamethasone; Calcium Dobesilate; Dexrazoxane; Doxorubicin; Etoposide; Hydrocortisone; Leucovorin; Mercaptopurine; Methotrexate; nelarabine; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Initial Low Risk (Initial LR) (Other): Meets all the following criteria: B-ALL, Age 1-<15 years, WBC < 50,000/microliter, CNS-1 or CNS-2, no BCR-ABL1, no iAMP21, and no VHR characteristics.
  Treated with Induction IA (vincristine, dexamethasone, pegaspargase), Induction IB (cyclophosphamide, cytarabine, mercaptopurine), Consolidation IA (vincristine, high-dose methotrexate + leucovorin, mercaptopurine). IT chemotherapy in all phases. Final risk group assigned by end of Consolidation IA.
  Interventions: Drug: Pegaspargase; Drug: Erwinia asparaginase; Drug: Cyclophosphamide; Drug: CYTARABINE; Drug: DEXAMETHASONE; Drug: HYDROCORTISONE; Drug: LEUCOVORIN CALCIUM; Drug: MERCAPTOPURINE; Drug: METHOTREXATE; Drug: Vincristine
- Initial High Risk (Initial HR) (Other): Meets at least one of the following criteria: Age >=15 years, WBC >=50,000/microliter, CNS-3, T-ALL, iAMP21, BCR-ABL1
  And: No VHR characteristics
  Treated with Induction IA (vincristine, dexamethasone, pegaspargase, doxorubicin + dexrazoxane), Induction IB (cyclophosphamide, cytarabine, mercaptopurine), Consolidation IA (vincristine, high-dose methotrexate + leucovorin, mercaptopurine). IT chemotherapy in all phases. Final risk group assigned by end of Consolidation IA.
  Interventions: Drug: Pegaspargase; Drug: Erwinia asparaginase; Drug: Cyclophosphamide; Drug: CYTARABINE; Drug: DEXAMETHASONE; Drug: Dexrazoxane; Drug: Doxorubicin; Drug: HYDROCORTISONE; Drug: LEUCOVORIN CALCIUM; Drug: MERCAPTOPURINE; Drug: METHOTREXATE; Drug: Vincristine
- Initial Very High Risk (Initial VHR) (Other): Any of the following are present: IKZF1 deletion, MLL (KMT2A) rearrangement, low hypodiploidy, t(17;19)
  Treated with Induction IA (vincristine, dexamethasone, pegaspargase, doxorubicin + dexrazoxane), Induction IB (cyclophosphamide, cytarabine, mercaptopurine), Consolidation IA (vincristine, high-dose methotrexate + leucovorin, mercaptopurine). IT chemotherapy in all phases. Final risk group assigned by end of Consolidation IA.
  Interventions: Drug: Pegaspargase; Drug: Erwinia asparaginase; Drug: Cyclophosphamide; Drug: CYTARABINE; Drug: DASATINIB; Drug: DEXAMETHASONE; Drug: Dexrazoxane; Drug: Doxorubicin; Drug: ETOPOSIDE; Drug: HYDROCORTISONE; Drug: LEUCOVORIN CALCIUM; Drug: MERCAPTOPURINE; Drug: METHOTREXATE; Drug: NELARABINE; Drug: Vincristine
- Final Low Risk (Final LR) (Other): Initial Low Risk and Low MRD (<0.0001) at first time point (Day 32)
  Final Risk Group assigned at end of Consolidation IA. Subsequent therapy as follows:
  CNS phase (vincristine, dexamethasone, mercaptopurine, pegaspargase [by randomization or direct assignment], IT chemotherapy); Consolidation II (vincristine, dexamethasone, mercaptopurine, methotrexate, pegaspargase [by randomization or direct assignment], IT chemotherapy); Continuation (vincristine, dexamethasone, mercaptopurine, methotrexate, IT chemotherapy).
  All treatment completed 24 months from date of complete remission.
  Interventions: Drug: Pegaspargase; Drug: Erwinia asparaginase; Drug: CYTARABINE; Drug: DEXAMETHASONE; Drug: HYDROCORTISONE; Drug: MERCAPTOPURINE; Drug: METHOTREXATE; Drug: Vincristine
- Final Intermediate Risk (Final IR) (Other): Initial High Risk and Low MRD (<0.0001) at first time point (Day 32)
  Final Risk Group assigned at end of Consolidation IA. Subsequent therapy as follows:
  CNS phase (vincristine, dexamethasone, mercaptopurine, pegaspargase [by randomization or direct assignment], IT chemotherapy); Consolidation II (vincristine, dexamethasone, mercaptopurine, doxorubicin + dexrazoxane, pegaspargase [by randomization or direct assignment], IT chemotherapy); Continuation (vincristine, dexamethasone, mercaptopurine, methotrexate, IT chemotherapy).
  All treatment completed 24 months from date of complete remission.
  Interventions: Drug: Pegaspargase; Drug: Erwinia asparaginase; Drug: CYTARABINE; Drug: DEXAMETHASONE; Drug: Dexrazoxane; Drug: Doxorubicin; Drug: HYDROCORTISONE; Drug: MERCAPTOPURINE; Drug: METHOTREXATE; Drug: Vincristine
- Final High Risk (Final HR) (Other): Initial Low Risk or Initial High Risk with High MRD (>=0.0001) at first time point (Day 32) but low MRD (<0.001) at second time point (week 10-12)
  Final Risk Group assigned at end of Consolidation IA. Subsequent therapy as follows:
  CNS phase (vincristine, dexamethasone, mercaptopurine, pegaspargase [by randomization or direct assignment], IT chemotherapy); Consolidation II (vincristine, dexamethasone, mercaptopurine, doxorubicin + dexrazoxane, pegaspargase [by randomization or direct assignment], IT chemotherapy); Continuation (vincristine, dexamethasone, mercaptopurine, methotrexate, IT chemotherapy).
  All treatment completed 24 months from date of complete remission.
  Interventions: Drug: Pegaspargase; Drug: Erwinia asparaginase; Drug: CYTARABINE; Drug: DEXAMETHASONE; Drug: Dexrazoxane; Drug: Doxorubicin; Drug: HYDROCORTISONE; Drug: MERCAPTOPURINE; Drug: METHOTREXATE; Drug: Vincristine
- Final Very High Risk (Final VHR) (Other): Initial VHR or any patient with high MRD (>=0.001) at second time point (week 10-12)
  Final Risk Group assigned at end of Consolidation IA. Subsequent therapy as follows:
  Consolidation IB/B-ALL (High-dose methotrexate + leucovorin, cyclophosphamide, etoposide, IT chemotherapy); Consolidation IB/T-ALL (nelararbine, cyclophosphamide, etoposide); Consolidation IC (High-dose cytarabine, etoposide, dexamethasone, pegaspargase [by direct assignment], IT chemotherapy); CNS phase (vincristine, dexamethasone, mercaptopurine, pegaspargase [by direct assignment], IT chemotherapy); Consolidation II (vincristine, dexamethasone, mercaptopurine, doxorubicin + dexrazoxane, pegaspargase [by direct assignment], IT chemotherapy); Continuation (vincristine, dexamethasone, mercaptopurine, methotrexate, IT chemotherapy).
  Dasatinib administered daily during all phases to pts with ABL1-class fusions. All treatment completed 24 months from date of complete remission.
  Interventions: Drug: Pegaspargase; Drug: Erwinia asparaginase; Drug: Cyclophosphamide; Drug: CYTARABINE; Drug: DASATINIB; Drug: DEXAMETHASONE; Drug: Dexrazoxane; Drug: Doxorubicin; Drug: ETOPOSIDE; Drug: HYDROCORTISONE; Drug: LEUCOVORIN CALCIUM; Drug: MERCAPTOPURINE; Drug: METHOTREXATE; Drug: NELARABINE; Drug: Vincristine
- Fixed Dose Pegaspargase (Active Comparator): Final LR, IR, HR patients who consent to randomization and are assigned to receive 15 doses of pegaspargase every 2-weeks at standard fixed-dose (2500 IU/m2/dose).
  Interventions: Drug: Pegaspargase; Drug: Erwinia asparaginase
- Reduced Dose (PK-Adjusted) Pegaspargase (Experimental): Final LR, IR, HR patients who consent to randomization and are assigned to receive 15 doses of pegaspargase every 2-weeks beginning at a reduced dose (2000 IU/m2/dose); subsequent doses adjusted based on nadir serum asparaginase activity (NSAA) levels, with goal of maintaining NSAA between 0.4 and 1.0 IU/mL. Closed to Enrollment.
  Interventions: Drug: Pegaspargase; Drug: Erwinia asparaginase
- Direct Assignment (Other): All VHR patients, and any Final LR, IR, HR patients who decline randomization: Assigned to receive standard dosing of pegaspargase (15 doses of pegaspargase every 2-weeks at standard fixed-dose; 2500 IU/m2/dose).
  Interventions: Drug: Pegaspargase; Drug: Erwinia asparaginase

INTERVENTIONS:
Drug: Pegaspargase — Arm A: Standard/Fixed Dose Pegaspargase (2500 IU/m2 every 2 weeks) Arm B: Reduced Dose (PK-adjusted) Pegaspargase (Starting Dose: 2000 IU/m2) Arm X: Directly Assigned Standard Dose (2500 IU/m2): For all VHR and patients who decline randomization
Drug: Erwinia asparaginase — Only for patients with Pegaspargase allergy or silent inactivation.
  Other Names: ERWINAZE®; ERWINIA CHRYSANTHEMI; ERWINASE®
Drug: Cyclophosphamide — Standard of Care
  Other Names: CYTOXAN
  Arms: Final Very High Risk (Final VHR); Initial High Risk (Initial HR); Initial Low Risk (Initial LR); Initial Very High Risk (Initial VHR)
Drug: CYTARABINE — Standard of Care
  Other Names: CYTOSINE ARABINOSIDE; ARA-C; CYTOSAR®
  Arms: Final High Risk (Final HR); Final Intermediate Risk (Final IR); Final Low Risk (Final LR); Final Very High Risk (Final VHR); Initial High Risk (Initial HR); Initial Low Risk (Initial LR); Initial Very High Risk (Initial VHR)
Drug: DASATINIB — Standard of Care
  Arms: Final Very High Risk (Final VHR); Initial Very High Risk (Initial VHR)
Drug: DEXAMETHASONE — Standard of Care
  Other Names: DECADRON®; HEXADROL®,; DEXONE®,; DEXAMETH®
  Arms: Final High Risk (Final HR); Final Intermediate Risk (Final IR); Final Low Risk (Final LR); Final Very High Risk (Final VHR); Initial High Risk (Initial HR); Initial Low Risk (Initial LR); Initial Very High Risk (Initial VHR)
Drug: Dexrazoxane — Standard of Care
  Other Names: Zinecard
  Arms: Final High Risk (Final HR); Final Intermediate Risk (Final IR); Final Very High Risk (Final VHR); Initial High Risk (Initial HR); Initial Very High Risk (Initial VHR)
Drug: Doxorubicin — Standard of Care
  Other Names: ADRIAMYCIN®
  Arms: Final High Risk (Final HR); Final Intermediate Risk (Final IR); Final Very High Risk (Final VHR); Initial High Risk (Initial HR); Initial Very High Risk (Initial VHR)
Drug: ETOPOSIDE — Standard of Care
  Other Names: VePesid
  Arms: Final Very High Risk (Final VHR); Initial Very High Risk (Initial VHR)
Drug: HYDROCORTISONE — Standard of Care
  Arms: Final High Risk (Final HR); Final Intermediate Risk (Final IR); Final Low Risk (Final LR); Final Very High Risk (Final VHR); Initial High Risk (Initial HR); Initial Low Risk (Initial LR); Initial Very High Risk (Initial VHR)
Drug: LEUCOVORIN CALCIUM — Standard of Care
  Arms: Final Very High Risk (Final VHR); Initial High Risk (Initial HR); Initial Low Risk (Initial LR); Initial Very High Risk (Initial VHR)
Drug: MERCAPTOPURINE — Standard of Care
  Other Names: 6-MP
  Arms: Final High Risk (Final HR); Final Intermediate Risk (Final IR); Final Low Risk (Final LR); Final Very High Risk (Final VHR); Initial High Risk (Initial HR); Initial Low Risk (Initial LR); Initial Very High Risk (Initial VHR)
Drug: METHOTREXATE — Standard of Care
  Arms: Final High Risk (Final HR); Final Intermediate Risk (Final IR); Final Low Risk (Final LR); Final Very High Risk (Final VHR); Initial High Risk (Initial HR); Initial Low Risk (Initial LR); Initial Very High Risk (Initial VHR)
Drug: NELARABINE — Standard of Care
  Arms: Final Very High Risk (Final VHR); Initial Very High Risk (Initial VHR)
Drug: Vincristine — Standard of Care
  Other Names: Oncovin
  Arms: Final High Risk (Final HR); Final Intermediate Risk (Final IR); Final Low Risk (Final LR); Final Very High Risk (Final VHR); Initial High Risk (Initial HR); Initial Low Risk (Initial LR); Initial Very High Risk (Initial VHR)

SUMMARY:
Acute lymphoblastic leukemia (ALL) is the most common cancer diagnosed in children. The cancer comes from a cell in the blood called a lymphocyte. Normal lymphocytes are produced in the bone marrow (along with other blood cells) and help fight infections. In ALL, the cancerous lymphocytes are called lymphoblasts. They do not help fight infection and crowd out the normal blood cells in the bone marrow so that the body cannot make enough normal blood cells. ALL is always fatal if it is not treated. With current treatments, most children and adolescents with this disease will be cured.

The standard treatment for ALL involves about 2 years of chemotherapy. The drugs that are used, and the doses of the drugs, are similar but not identical for all children and adolescents with ALL. Some children and adolescents receive stronger treatment, especially during the first several months. A number of factors are used to decide how strong the treatment should be to give the best chance for cure. These factors are called "risk factors". This trial is studying the use of a new, updated set of risk factors to decide how strong the treatment will be. The study also will test a new way of dosing a chemotherapy drug called pegaspargase (which is part of the standard treatment for ALL) based on checking levels of the drug in the blood and adjusting the dose based on the levels.

DETAILED DESCRIPTION:
There are a standard set of risk factors which are used to decide how strong treatment should be for a child with ALL. These risk factors include the child's age when the leukemia is diagnosed, how high the white blood cell count (WBC) is in the blood, whether or not leukemia cells are seen in the spinal fluid (referred to as Central Nervous System or CNS status), and whether or not the leukemia has certain abnormalities in their chromosomes (genetic material in the cell). Another risk factor is the amount of leukemia in the marrow that can be measured by a special laboratory test called "MRD" (Minimal Residual Disease) after the first month of treatment.

Over the last several years, new factors have been identified which help predict how well a child's leukemia may respond to treatment. These new risk factors include additional abnormalities in the genes of the leukemia cell, as well the amount of leukemia (MRD level) at second time point (about 2-3 months after starting treatment).

In this trial, the investigators will use the new risk factors along with old risk factors to decide how strong the treatment will be. The goal is to better identify those participants who might benefit from stronger treatment in order to improve their chance for cure. The investigators also hope to better identify participants who have a high chance of being cured with standard treatment in order to reduce their chance of side effects while maintaining the chance of cure.

This trial also aims to study the dosing of a drug called pegaspargase. Pegaspargase is a chemotherapy drug that is an important part of ALL treatment but it is also can cause many side effects. With the standard dose of pegaspargase, levels of the drug in the blood are higher than may be necessary to effectively treat leukemia.

On this research study, the investigators will be comparing the standard dose of pegaspargase with a new way of dosing the drug based on levels of the drug that we can measure in the blood. With the new way of doing, treatment will begin with a lower dose. If the levels are high, the dose will be decreased one more time; however, if at any time the levels are too low, dosing will be switched back up to the standard dose. The goal of this research study is to learn whether this new way of dosing (starting at a lower dose and changing the dose based on drug levels in the blood) will decrease side effects but still be as effective as the standard dosing of the drug.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of acute lymphoblastic leukemia. Diagnosis should be made by bone marrow aspirate or biopsy demonstrating ≥ 25% involvement by lymphoblasts, with flow cytometry or immunohistochemistry confirming B-precursor or T-ALL phenotype.

   -- For patients with circulating blasts in the peripheral blood, flow cytometry confirmation of B-ALL or T-ALL phenotype is sufficient for registration onto the study. Bone marrow aspirate and/or biopsy should be performed as soon as feasible, preferably prior to the initiation of any therapy.
2. Prior Therapy: No prior therapy is allowed except for the following:

   * Corticosteroids: Short courses of corticosteroid (defined as ≤ 7 days of corticosteroids within the 4-weeks preceding registration) are allowed prior to registration.

     --- Participants who have been on corticosteroids chronically (defined as more than 7 days of corticosteroids within the 4-weeks preceding registration or more than 28 days of corticosteroids over the preceding 6 months) are not eligible.
   * IT cytarabine: A single dose of intrathecal cytarabine (at the time of the diagnostic lumbar puncture) is allowed prior to registration. If patient has received IT cytarabine prior to registration, Day 1 IT cytarabine should not be administered.
   * Emergent Radiation Therapy: Emergent radiation to the mediastinum or other life-threatening masses is allowed prior to registration.
3. Age: 365 days to < 22 years
4. Direct bilirubin < 1.4 mg/dL (23.9 micromoles/L).
5. Ability of parent or guardian to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Mature B-cell (Burkitt's) ALL (defined by the presence of surface immunoglobulin and/or the t(8;14)(q24;q32), t(8;22), or t(2;8) translocation and/or c-myc-gene rearrangement).
2. World Health Organization diagnostic criteria of mixed phenotype acute leukemia (MPAL) or leukemia of ambiguous lineage
3. Any chemotherapy or radiotherapy for previous malignancy are not eligible.
4. Treatment in past with any anti-neoplastic agent, including methotrexate, 6-mercaptopurine, 6-thioguanine, vincristine cyclophosphamide, cytarabine (except for IT cytarabine), or any anthracycline, for any reason (eg, rheumatologic or autoimmune condition).
5. Currently receiving any investigational agents.
6. Known HIV-positivity
7. Uncontrolled intercurrent illness including, but not limited to ongoing infection with vital sign instability (hypotension, respiratory insufficiency), life-threatening acute tumor lysis syndrome (eg, with renal failure), symptomatic congestive heart failure, cardiac arrhythmia, intracranial or other uncontrolled bleeding, or psychiatric illness/social situations that would limit compliance with study requirements.
8. Pregnant women are excluded from this study because many of the agents used on this protocol have potential for teratogenic and/or abortifacient effects. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with these chemotherapy agents, breastfeeding should be discontinued if the mother is enrolled.
9. History of a previous malignancy. Exception: Individuals with a previous malignancy treated with surgery only (no chemotherapy or radiotherapy) more than 5 years prior to registration may be enrolled.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 560 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2034-11 (Estimated)

PRIMARY OUTCOMES:
Complete Remission Rate | After 1 month of treatment (Induction IA) for all participants, assessed at the end of first month of treatment in all participants through study completion (expected to take 4-5 years to accrue)
Event-Free Survival | From registration to the time of induction failure, relapse, death, or second malignancy, whichever came first, assessed up to 60 months.

SECONDARY OUTCOMES:
Overall Survival | From registration to the time of death from any cause, assessed up to 60 months.
Disease Free Survival | From randomization or direct assignment (for participants who achieved a complete remission and were assigned a final risk group) to the time of relapse, death, or second malignancy, whichever came first, assessed up to 60 months.
Nadir Serum Asparaginase Activity (NSAA) | During post-induction therapy with 30-weeks of pegaspargase (15 doses), collected during the first 6 months of therapy for all participants through study completion (expected to take 4-5 years to accrue)
  Proportion of patients receiving pegaspargase with NSAA >= 1.0 IU/mL
Non-allergic Asparaginase Toxicity | During post-induction therapy with 30-weeks of pegaspargase (15 doses). collected during the first 6 months of therapy for all participants through study completion (expected to take 4-5 years to accrue)
  Frequency of non-allergic asparaginase-related toxicities, an average of 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Burns, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (9):
- United States (7):
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Columbia University Medical Center, Morgan Stanley Children's Hospital of New York-Presbyterian, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Hasbro Children's Hospital / Rhode Island Hospital, Providence, Rhode Island
- Canada (2):
  - Hospital Sainte Justine, University of Montreal, Montreal, Quebec
  - Centre Hospitalier U. de Quebec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park Y, K C N, Willekens J, Patel C, Savage BA, Lin H, Paneque A, Daly R, Thrope A, Burns MA, Welch JJG, Kahn JM, Kelly KM, Tran TH, Michon B, Gennarini L, Silverman LB, Sands SA, Cole PD. Treatment-Related Changes in Cerebrospinal Fluid Markers of Oxidative Stress and Neurodegeneration during Therapy for Childhood Acute Lymphoblastic Leukemia. Cancer Epidemiol Biomarkers Prev. 2025 Nov 3;34(11):2015-2024. doi: 10.1158/1055-9965.EPI-25-1058. PMID 40905823
- [Derived] Tran TH, Langlois S, Meloche C, Caron M, Saint-Onge P, Rouette A, Bataille AR, Jimenez-Cortes C, Sontag T, Bittencourt H, Laverdiere C, Lavallee VP, Leclerc JM, Cole PD, Gennarini LM, Kahn JM, Kelly KM, Michon B, Santiago R, Stevenson KE, Welch JJG, Schroeder KM, Koch V, Cellot S, Silverman LB, Sinnett D. Whole-transcriptome analysis in acute lymphoblastic leukemia: a report from the DFCI ALL Consortium Protocol 16-001. Blood Adv. 2022 Feb 22;6(4):1329-1341. doi: 10.1182/bloodadvances.2021005634. PMID 34933343